CLINICAL TRIAL: NCT06356168
Title: Social Virtual Reality to Alleviate Loneliness and Symptoms for Individuals Receiving Hemodialysis
Brief Title: Virtual Reality in End Stage Kidney Disease
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SVR/IVR
Record Dates: First submitted 2024-03-28; First posted 2024-04-10 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: End Stage Kidney Disease
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Social Virtual Reality (Experimental): Social Virtual Reality will be delivered using virtual reality glasses for 30-45 minutes during dialysis sessions. Groups of 3 participants will watch a movie or program together through the glasses. They will be able to talk and interact during the session.
  Interventions: Behavioral: Social Virtual Reality
- Individual Virtual Reality (Active Comparator): Individual Virtual Reality will be delivered using virtual reality glasses for 30-45 minutes during dialysis sessions. Those randomized to this arm will watch a movie or program alone through the glasses.
  Interventions: Behavioral: Individual Virtual Reality

INTERVENTIONS:
Behavioral: Social Virtual Reality — Participants interact using virtual reality during dialysis.
  Arms: Social Virtual Reality
Behavioral: Individual Virtual Reality — Participants use virtual reality alone during dialysis.
  Arms: Individual Virtual Reality

SUMMARY:
The goal of this clinical trial to compare the social virtual reality and individual virtual reality in patients with end stage kidney disease who are hemodialysis. The main aim is to determine if there are differences in symptoms between the groups. Participants will use virtual reality glasses for 30-45 minutes during dialysis sessions for 4 weeks.

DETAILED DESCRIPTION:
In a single site, 2-arm (Social Virtual Reality group; Individual Virtual Reality Group), parallel, randomized controlled trial we will enroll 60 subjects (n=30 per group) to assess the effects of Social Virtual Reality to Individual Virtual Reality on symptoms in participants with end stage kidney disease who are receiving hemodialysis.

To compare the effects of social virtual reality to individual virtual reality on loneliness To explore the effects of social virtual reality to individual virtual reality on anxiety and depression.

To compare the effects social virtual reality to individual virtual reality on quality of life.

ELIGIBILITY:
Inclusion Criteria

* Diagnosis of end stage kidney disease with hemodialysis 3 times per week for at least 1 month

Exclusion Criteria

* Acutely ill
* Active nausea
* Epilepsy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
De Jong Gierveld Scale | Baseline and 4 Weeks
  Measures how bad or severe a person's loneliness is. Score range from 11-44; higher scores indicate more loneliness.

CONTACTS AND LOCATIONS:
Overall Officials: Lea Ann Matura, PhD, Principal Investigator — University of Pennsylvania

IPD SHARING:
Plan to Share IPD: No